CLINICAL TRIAL: NCT06622655
Title: Agilik@Home: Demonstrate the Clinical Improvement Due to the Home Use of Agilik in Children With Cerebral Palsy
Brief Title: Clinical Improvement Due to the Home Use of Agilik in Children With Cerebral Palsy
Acronym: Agilik@home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: IRCCS Fondazione Stella Maris (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Fondazione Mondino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIP1122; PNC0000007 (Other Grant/Funding Number: Italian Ministry of Research)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy (CP)
Keywords: exoskeleton device; powered orthosis; cerebral palsy; crouch gait; home use
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Home rehabilitation
  Interventions: Device: Powered orthosis
- Control Group (No Intervention)

INTERVENTIONS:
Device: Powered orthosis — Home rehabilitation (2 months, 30 minutes/day, 5 days/week) during which subjects will practice walking with the device at home.
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to learn if a two month training with the Agilik powered orthosis improves the knee extension or the endurance in pediatric patients with Cerebral palsy and a crouch gait. It will also learn about the safety of Agilik. The main questions it aims to answer are:

Does the Agilik powered orthosis increase the value of the knee extension during walking? What medical problems do participants have when using the Agilik powered orthosis? Researchers will compare a group of patients using the Agilik powered exoskeleton with a group of patients treated with standard therapy.

Participants will:

Use Agilik at home or perform standard therapy for 2 months Visit the clinic at the beginning of the study, after 3 months and after 1 additional month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP and a crouch gait
* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study, or alternatively, ability to do so based on parent report and physician observation during history and physical examination.
* Body weight between 20 and 125 Kg
* Knee flexion retraction assessed in supine position by less than 10°. Hamstring contracture as assessed by straight leg raising test does not limit ability to participate in the study.
* Subjects must not have had a tibio-tarsal arthrodesis. In addition, they must have at least 5° of passive dorsi-flexion of the ankle.
* Able to walk at least 3 m without stopping, with or without a walking aid.
* Able to understand and follow simple directions based on parent report and physician observation during historical and physical examination.
* GMFCS level I, II and III
* MAS score ≤ 2

Exclusion Criteria:

* Any severe neurological, musculoskeletal and/or cardiorespiratory involvement preventing the ability to walk;
* A history of uncontrolled seizure in the past year
* Severe spasticity
* Hip and/or knee flexion contracture of more than 20°

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Endurance | Baseline, 3 months and 4 months
  Distance walked during a 6-minutes walking test (6MWT)
Knee extension in mid stance (KEMS) | Baseline, 3 months and 4 months
  Anti-gravity knee extension in mid stance measured with quantitative gait analysis

SECONDARY OUTCOMES:
Measurements of the Joint range of motions (ROMs) and muscle lengths | Baseline, 3 months and 4 months
  Joint Range of motions and muscle lengths as measured by therapists
Level of spasticity in the lower limbs | Baseline, 3 months and 4 months
  Assessed with the Modified Ashworth scale (MAS)
Walking speed | Baseline, 3 months and 4 months
  Assessed with the 10-meter walking test (10mWT)
Postural and motor abilities | Baseline, 3 months and 4 months
  Assessed with the Gross Motor Function Measure-88 (GMFM-88)
Gait pattern | Baseline, 3 months and 4 months
  Assessed with overground 3D gait analysis with electromyography (EMG) data acquisition
Self-perception of performance in everyday living | Baseline, 3 months and 4 months
  Assessed with the Canadian Occupational Performance Measure (COPM)
Static balance | Baseline, 3 months and 4 months
  Assessed with Centre of Pressure (COP) detection using the force platforms of the gait analysis.
Usability and acceptability of the powered orthosis | After the treatment only in the intervention group
  Assessed with the System Usability Scale (SUS) and the Technology Acceptance Method 3 (TAM-3)
Behavioural engagement | After the treatment only in the intervention group
  Assessed with semi-structured interviews

OTHER OUTCOMES:
Spatiotemporal parameters of gait during daily life | Between baseline and month 3
  Remote monitoring of gait behavior assessed with sensorized shoes

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - IRCCS E. MEDEA - Associazione "La Nostra Famiglia", Bosisio Parini, Lecco
  - IRCCS Fondazione Stella Maris, Calambrone, Pisa
  - Fondazione Don Carlo Gnocchi Onlus - IRCCS S. Maria Nascente, Milan
  - Fondazione Mondino, Pavia
  - Fondazione Don Carlo Gnocchi Onlus, Roma
  - Fondazione Don Carlo Gnocchi Onlus - Centro S. Maria al Mare, Salerno

IPD SHARING:
Plan to Share IPD: Yes
The results obtained at the end of this clinical trial will be presented at national and international conferences and submitted to peer-reviewed international journals. The raw data of the study will be published among the supplementary materials of scientific articles and/or uploaded to Zenodo, a multidisciplinary repository, managed by CERN in Geneva, which allows researchers to share and preserve research results in any size and form. Depositing data in ZENODO guarantees their compliance with the FAIR principles.
Supporting Information: Study Protocol, SAP